CLINICAL TRIAL: NCT03759262
Title: Pilot Study of Transplant-related Events in Patients Receiving Ultra-high-dose Vitamin D Supplementation
Brief Title: Ultra-high Dose Vitamin D for HSCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Etan Orgel, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-18-00362
Record Dates: First submitted 2018-11-08; First posted 2018-11-29 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: vitamin D; cytokines
MeSH Terms: interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vitamin D (Cholecalciferol) (Experimental): All subjects will be enrolled to this arm. A single dose of ultra-high-dose vitamin D will be given.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — A single dose of ultra-high-dose vitamin D (cholecalciferol) will be given prior to hematopoietic stem cell transplant. Research labs including inflammatory biomarker panels will be obtained prior to and after the dose is given.
  Other Names: vitamin D

SUMMARY:
This is a pilot study to investigate the effects of achieving adequate vitamin D levels via ultra-high-dose vitamin D supplementation given prior to hematopoietic stem cell transplant on transplant-related complications and inflammatory biomarkers.

DETAILED DESCRIPTION:
Up to 70% of patients have vitamin D deficiency prior to hematopoietic stem cell transplant (HSCT). Patients with sufficient Vitamin D levels (>50nm/L) prior to allogeneic transplant have significantly better overall survival (OS) and lower rates of rejection and relapse. Vitamin D inhibits Th1 and augments Th2 cell development. Patients who receive vitamin D supplementation during allogeneic transplant have less inflammatory-mediated processes such as chronic graft versus host disease (GVHD) and lower levels of naïve CD8+ cells and CD40 ligand. Multiple studies have raised concern regarding the adequacy of standard and high-dose vitamin D dosing for vitamin D deficiency. A single oral ultra-high dose of Vitamin D given prior to HSCT has been shown to be a safe and well tolerated method of sustaining therapeutic Vitamin D levels for 6-19 weeks.

This is a pilot study to investigate the dynamic changes in inflammatory biomarkers following ultra-high-dose vitamin D supplementation. The study population is patients with total vitamin D level </=50ng/mL prior to HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are preparing for HSCT
* If a patient is receiving an autologous transplant, enrollment must occur prior to first transplant in the case that the patient is planned for multiple transplants

Exclusion Criteria:

* Uncorrected hypocalcemia or hypophosphatemia
* Patients in the ICU or on renal replacement therapy
* Patients who have had an allogeneic transplant within the past 12 months prior to enrollment

Enrolled patients with 25OHD level ≤50 ng/mL continue on study

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Incidence of graft-versus-host disease, veno-occlusive disease, and thrombotic microangiopathy | 100 days after transplant
  Graft-versus-host disease, veno-occlusive disease, and thrombotic microangiopathy
Vitamin D sufficiency following Stoss dosing | prior to transplant
  Vitamin D sufficiency following Stoss dosing prior to tranpslantation

SECONDARY OUTCOMES:
Rates of survival, relapse, and significant infections | from time of transplant to 1 year after transplant
  Clinically significant events including but not limited to survival, relapse, significant infections.
Cytokine levels | before vitamin D is given, 1-2 weeks after vitamin D is given, day of transplant, day +7, day +14, and day +30
  The investigators will examine changes in levels of IFN-gamma, TNF-alpha, IL-1a, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10 (in pg/mL) before and after vitamin D is given
Cytokine stimulation test | before vitamin D is given, and 1-2 weeks after vitamin D is given
  The investigators will examine changes in the immune profile (reactivity of CD45, 235, 61, 66 197, 19, 4, 38, 163, 43, 7, 62L, 127, 123, 279, 274, 14, 90, 11c, 294, 15, 16, 25, 27, 8, 33, 3, 45RA, 56, 11b; pS6, p-p38, HLA-DR, pERK 1/2, pStat3, pStat1, TCRgd, pStat5) in response to cytokine stimulation before and after vitamin D is given

CONTACTS AND LOCATIONS:
Overall Officials: Etan Orgel, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallace G, Jodele S, Howell J, Myers KC, Teusink A, Zhao X, Setchell K, Holtzapfel C, Lane A, Taggart C, Laskin BL, Davies SM. Vitamin D Deficiency and Survival in Children after Hematopoietic Stem Cell Transplant. Biol Blood Marrow Transplant. 2015 Sep;21(9):1627-31. doi: 10.1016/j.bbmt.2015.06.009. Epub 2015 Jun 18. PMID 26093045
- [Background] Wallace G, Jodele S, Myers KC, Dandoy CE, El-Bietar J, Nelson A, Teusink-Cross A, Khandelwal P, Taggart C, Gordon CM, Davies SM, Howell JC. Single Ultra-High-Dose Cholecalciferol to Prevent Vitamin D Deficiency in Pediatric Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2018 Sep;24(9):1856-1860. doi: 10.1016/j.bbmt.2018.05.019. Epub 2018 May 18. PMID 29782992
- [Background] Hansson ME, Norlin AC, Omazic B, Wikstrom AC, Bergman P, Winiarski J, Remberger M, Sundin M. Vitamin d levels affect outcome in pediatric hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2014 Oct;20(10):1537-43. doi: 10.1016/j.bbmt.2014.05.030. Epub 2014 Jun 5. PMID 24910378
- [Background] Caballero-Velazquez T, Montero I, Sanchez-Guijo F, Parody R, Saldana R, Valcarcel D, Lopez-Godino O, Ferra I Coll C, Cuesta M, Carrillo-Vico A, Sanchez-Abarca LI, Lopez-Corral L, Marquez-Malaver FJ, Perez-Simon JA; GETH (Grupo Espanol de Trasplante Hematopoyetico). Immunomodulatory Effect of Vitamin D after Allogeneic Stem Cell Transplantation: Results of a Prospective Multicenter Clinical Trial. Clin Cancer Res. 2016 Dec 1;22(23):5673-5681. doi: 10.1158/1078-0432.CCR-16-0238. Epub 2016 Jun 29. PMID 27358490
- [Background] van Etten E, Mathieu C. Immunoregulation by 1,25-dihydroxyvitamin D3: basic concepts. J Steroid Biochem Mol Biol. 2005 Oct;97(1-2):93-101. doi: 10.1016/j.jsbmb.2005.06.002. Epub 2005 Jul 19. PMID 16046118